CLINICAL TRIAL: NCT05009238
Title: Effect of Lumbar Stabilization Exercises on Balance and Spatiotemporal Gait Parameters in Postmenopausal Women
Brief Title: Effect of l S Exercises on Balance and Spatiotemporal Gait Parameters in P M Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hend Hamdy (Other)
Responsible Party: Sponsor-Investigator, Hend Hamdy, lecturer of pt for basic science, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: p.T.RCE/012/003190
Record Dates: First submitted 2021-07-23; First posted 2021-08-17 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Postmenopausal

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Experimental): Group (A): will receive lumbar stabilization exercises
  Interventions: Other: lumbar stabilization exercises
- Group (B) (No Intervention): Group (B): will be control group.

INTERVENTIONS:
Other: lumbar stabilization exercises — selected exercises will taught to participant and practiced 3 times per week for 6 weeks
  Arms: Group (A)

SUMMARY:
Menopause is a natural process in women's life with hormonal fluctuations that cause physical and emotional symptoms such as(Hot flashes, insomnia, physical in activity, unstable mood, difficulties in memory and concentration, anxiety, stress, irritability, unstable body mass, sexual dysfunction, feelings of sadness, infertility, and depression).

Balance disturbances are common in the community as a whole and increase in frequency with age. The risk of falling increases from age 45 in women and peaks in the 55-59-year age group. Around the time of the menopause, estrogen production decreases dramatically and bone loss accelerates, which predisposes for fractures if a fall occurs.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women: Their age will be ranged between 45-59 years old, with low back pain.

Exclusion Criteria:

* Infection disease or fever.
* Foot ulcers.
* Foot infection or undergoing foot surgery.
* Recent fracture in foot and toes with unhealed wounds.
* Thrombotic disease of lower extremities.
* Deep proprioception loss.
* Peripheral neuropathy.
* Gout or advanced arthritis affecting the foot and toes.

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Step length | about 6 weeks.
  the distance between the point of initial contact of one foot and the point of initial contact of the opposite foot measured by cm
step symmetry | about 6 weeks.
  right to left time distribution measured by second
walking speed | about 6 weeks.
  the ratio of distance to the time in which the distance was covered by the subject measured by m/s

IPD SHARING:
Plan to Share IPD: Yes